CLINICAL TRIAL: NCT03366597
Title: Effect of Sevoflurane on the Content of S100β in Infants With Congenital Heart Disease Undergo Cardiac Surgery.
Brief Title: The Research of the Effect of Sevoflurane on Brain-protection of Cardiac Surgery in Infants.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Ma (Other)
Responsible Party: Sponsor-Investigator, Jun Ma, The Chief of Anesthesiology Department, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017030X
Record Dates: First submitted 2017-11-21; First posted 2017-12-08 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Congenital Heart Disease; Infant, Premature, Diseases
Keywords: sevoflurane; S100β protein; regional cerebral oxygen saturation; infant
MeSH Terms: conditions — Heart Defects, Congenital; Infant, Premature, Diseases | interventions — Sevoflurane

STUDY DESIGN:
Intervention Model Description: one group is treated with sevoflurane, the other is not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sevoflurane (Experimental): Sevoflurane will be used as a narcotic drug in one group during cardiac surgery.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — 1.5%-3% Sevoflurane will be given during the cardiac surgery except cardiopulmonary bypass.

SUMMARY:
To observe the effect of sevoflurane on the concentration of S100β and regional cerebral oxygen saturation in infants with congenital heart disease undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of congenital heart disease
* Undergoing heart surgery with cardiopulmonary bypass

Exclusion Criteria:

* Pulmonary arterial hypertension
* Sevoflurane allergy

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2021-12-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Concentration of S100β protein | 5 minutes after tracheal intubation; immediately after cardiopulmonary bypass; immediately after operation; 12 hours, 24 hours postoperative
  The concentration of S100β protein was performed using the electrochemiluminescence immunoassay.(Blood samples from patients were drawn from central intravenous.)

SECONDARY OUTCOMES:
Level of regional cerebral oxygen saturation(rScO2) | 5 minutes after tracheal intubation; immediately after cardiopulmonary bypass; immediately after operation; 12 hours, 24 hours postoperative
  The rScO2 was measured by using noninvasive near-infrared spectroscopy during cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Boqun Cui, M.D., Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Fenton KN, Freeman K, Glogowski K, Fogg S, Duncan KF. The significance of baseline cerebral oxygen saturation in children undergoing congenital heart surgery. Am J Surg. 2005 Aug;190(2):260-3. doi: 10.1016/j.amjsurg.2005.05.023. PMID 16023442
- [Background] Rezaei O, Pakdaman H, Gharehgozli K, Simani L, Vahedian-Azimi A, Asaadi S, Sahraei Z, Hajiesmaeili M. S100 B: A new concept in neurocritical care. Iran J Neurol. 2017 Apr 4;16(2):83-89. PMID 28761630
- [Background] Stojanovic Stipic S, Carev M, Bajic Z, Supe Domic D, Roje Z, Jukic A, Stipic T. Increase of plasma S100B and neuron-specific enolase in children following adenotonsillectomy: a prospective clinical trial. Eur Arch Otorhinolaryngol. 2017 Oct;274(10):3781-3788. doi: 10.1007/s00405-017-4698-1. Epub 2017 Aug 7. PMID 28785895
- [Background] Chen F, Duan G, Wu Z, Zuo Z, Li H. Comparison of the cerebroprotective effect of inhalation anaesthesia and total intravenous anaesthesia in patients undergoing cardiac surgery with cardiopulmonary bypass: a systematic review and meta-analysis. BMJ Open. 2017 Oct 11;7(10):e014629. doi: 10.1136/bmjopen-2016-014629. PMID 29025825
- [Background] Pironkova RP, Giamelli J, Seiden H, Parnell VA, Gruber D, Sison CP, Kowal C, Ojamaa K. Brain injury with systemic inflammation in newborns with congenital heart disease undergoing heart surgery. Exp Ther Med. 2017 Jul;14(1):228-238. doi: 10.3892/etm.2017.4493. Epub 2017 May 22. PMID 28672919